CLINICAL TRIAL: NCT00241436
Title: An Open-Label Pharmacokinetic and Pharmacodynamic Study of Anastrozole (Arimidex™) Used to Treat Pubertal Boys With Gynecomastia of Recent Onset
Brief Title: Open Label Arimidex in Gynecomastia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5394C00001
Record Dates: First submitted 2005-10-17; First posted 2005-10-19 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2011-01

CONDITIONS: Gynecomastia
MeSH Terms: conditions — Gynecomastia | interventions — Anastrozole

INTERVENTIONS:
Drug: Anastrozole (ARIMIDEX™)

SUMMARY:
The purpose of this study is to evaluate the safety, effectiveness, pharmacokinetics and pharmacodynamics of anastrozole (ARIMIDEX™) in the treatment of boys with gynecomastia.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent/assent (as per local requirements), males aged 11-18 yrs. (after his 10th and prior to 19th birthday), gynecomastia, one breast measuring ≥ 2 cm in diameter (by ultrasound or caliper measurement) that has not decreased during the prior 3 month period by medical history and has been present for 12 months or less (date of onset based on best estimate of treating physician after discussion with patient and or patient's parent/guardian), normal renal liver and thyroid function, no evidence of hormone producing tumor, no evidence of hypogonadism or androgen resistance.

Exclusion Criteria:

* Patients who have been given medications known to cause gynecomastia within the previous 6 months, involvement in the planning and conduct of the study (includes AZ staff and investigative site staff), previous enrollment in the present study, investigators opinion patient would be unable to comply with study protocol.

Ages: 11 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35
Dates: Start 2005-06; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Assess anastrazole PK in boys aged 11-18 yrs. in pubertal boys with gynecomastia of less than 12 months duration

SECONDARY OUTCOMES:
Determine efficacy by the response rate following 6 months of treatment

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Arimidex Medical Sciences Director, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Jacksonville, Florida, United States

REFERENCES:
- [Derived] Mauras N, Bishop K, Merinbaum D, Emeribe U, Agbo F, Lowe E. Pharmacokinetics and pharmacodynamics of anastrozole in pubertal boys with recent-onset gynecomastia. J Clin Endocrinol Metab. 2009 Aug;94(8):2975-8. doi: 10.1210/jc.2008-2527. Epub 2009 May 26. PMID 19470631